CLINICAL TRIAL: NCT07121985
Title: Multispectral Optoacoustic Imaging for the Detection of Inflammation and Damage of Peripheral Nerves in Guillain-Barré Syndrome and Chronic Inflammatory Demyelinating Polyneuropathy
Acronym: MIND
Status: Not yet recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, PD Dr. med. Dr. Humanbiol., University of Erlangen-Nürnberg Medical School
Other Study IDs: MIND_study
Record Dates: First submitted 2025-08-06; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: CIDP - Chronic Inflammatory Demyelinating Polyneuropathy; Guillain-Barré Syndrome (GBS)
Keywords: MSOT; PAI; Nerve Ultrasound
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Healthy Volunteers
- GBS patients: GBS patients
- CIDP patients: CIDP patients

SUMMARY:
The aim of this study is to assess disease activity in patients with Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) and Guillain-Barré Syndrome (GBS) using multispectral optoacoustic tomography (MSOT).

The currently available diagnostic procedures for CIDP and GBS do not allow for a clear distinction between remission and active disease and show limitations in sensitivity and specificity during acute diagnostics. This can lead to delayed diagnosis, which is crucial for timely initiation of therapy and, consequently, for a better prognosis. Long-term therapy management is also challenging, as objective parameters for assessing therapeutic success are largely lacking.

MSOT can detect inflammation through the measurement of hemoglobin, a method that our research group has already successfully demonstrated in patients with chronic inflammatory bowel diseases (Knieling, NEJM 2017). The use of MSOT could therefore also be applied to nerve inflammation, allowing for earlier detection of inflammation and nerve damage and contributing to timely treatment of patients.

For nerve imaging, a CE-certified MSOT device from iThera Medical is available at the Pediatric Clinic in Erlangen. In addition, a non-CE-certified device with lower laser power is available, which can be used for bedside examinations.

The arm nerves will be examined in three cohorts, which will be compared with each other and with standard diagnostics (blood tests, electrophysiology, conventional ultrasound).

Each cohort will include ten healthy control subjects, ten patients with CIDP, and ten patients with GBS.

ELIGIBILITY:
Inclusion Criteria Patient Cohort(s):

* Established diagnosis or suspected CIDP or GBS
* Age: 18 years or older
* Written informed consent provided by participant

Inclusion Criteria Control Cohort:

* Written informed consent provided by participant
* Age: 18 years or older
* No pre-existing conditions that may affect peripheral nerves (e.g., diabetes, traumatic nerve injuries, etc.)

Exclusion Criteria:

* Pregnancy
* Breastfeeding mothers
* Cardiopulmonary instability
* Tattoo in the examination area
* Subcutaneous fat tissue > 3 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Guillain-Barré Syndrome (GBS) and Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) are recruited from the Department of Neurology. All participants will have a confirmed diagnosis of GBS or CIDP based on established clinical and diagnostic criteria. Recruitment will occur during or following their routine clinical appointments. Eligible patients who provide informed consent will be invited to participate in the study assessments.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-08-06 (Estimated); Primary Completion 2026-08-06 (Estimated); Study Completion 2027-08-06 (Estimated)

PRIMARY OUTCOMES:
Single Wavelength PA signal | Single time point
  Photoacoustic single wavelength signal between 700nm and 1100nm in the measured nerves.
PA hemoglobin signal | Single time point
  Unmixed photoacoustic hemoglobin signal (oxygenated, deoxygenated and derived saturation) in the measured nerves
Doppler signal | Single time point
  Ultrasound-based Doppler signal in the measured nerves

SECONDARY OUTCOMES:
Nerve diameter | Single time point
  Ultrasound-based dimensional measurements of the respective nerve.
Clinical scores | Single time point
  Assessment of clinical scores (MRC, NIS) for correlation with imaging data.
PA lipid signal | Single time point
  Unmixed photoacoustic lipid signal in the measured nerves
PA water signal | Single time point
  Unmixed photoacoustic water signal in the measured nerves
PA collagen signal | Single time point
  Unmixed photoacoustic collagen signal in the measured nerves